CLINICAL TRIAL: NCT07057076
Title: The Role of Microbiome in Recurrence After Colorectal Cancer Surgery With Postoperative Organ/Space Surgical Site Infection
Brief Title: Microbiome and Colorectal Cancer Recurrence
Status: Completed | Type: Observational
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Blanca Montcusí Ventura, Colorectal Surgeon, Hospital del Mar
Other Study IDs: 2020/9513/I; PI19/00643 (Other Grant/Funding Number: Institute of Health Carlos III); SGR 00024 (Other Grant/Funding Number: Agency for Management of University and Research Grants (AGAUR))
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer Recurrent
Keywords: Colorectal cancer; Anastomotic leak; Microbiome; Tumor recurrence
MeSH Terms: conditions — Colorectal Neoplasms; Anastomotic Leak; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Peritoneal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colorectal cancer patients: Colorectal cancer patients operated on for cure and complicated by anastomotic leak

SUMMARY:
Anastomotic leak is associated with higher rates of tumor recurrence after colorectal cancer surgery. However, the mechanisms responsible remain unknown. The aim of this study is to identify associations between the peritoneal microbiome and recurrence in colorectal cancer patients with postoperative anastomotic leak. This is a single-center retrospective study of patients undergoing colorectal cancer surgery complicated with anastomotic leak between 2004 and 2012. Samples of peritoneal fluid were collected either through percutaneous drainage or reoperation, and microbiome was analyzed using whole genome shotgun. Oncological outcomes are registered. Associations between peritoneal microbiome and tumor recurrence are investigated.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer patients operated on for cure and complicated with anastomotic leak.

Exclusion Criteria:

* Non-curative resection.
* Urgent surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer patients operated on for cure and complicated with anastomotic leak.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Recurrence | 5 years
  Colorectal cancer recurrence after surgery

IPD SHARING:
Plan to Share IPD: No